CLINICAL TRIAL: NCT03440086
Title: Evaluation of One-hour Application of Abdominal Jackson-Pratt Drain in Order to Reduce Pain After Laparoscopic Surgery in Gynecology
Brief Title: Temporary Application of Abdominal Jackson-Pratt Drain to Reduce Pain After Laparoscopic Surgery in Gynecology
Acronym: DRAIN-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Medical Doctor, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DRAIN-1
Record Dates: First submitted 2018-02-06; First posted 2018-02-20 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain
Keywords: Laparoscopic surgery; Pain; Jackson-Pratt drain
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (no blinded)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Jackson-Pratt drain (Experimental): Patients in this arm will undergo one-hour application of abdominal Jackson-Pratt drain at the end of laparoscopic procedure.
  Interventions: Device: abdominal Jackson-Pratt drain
- Controls (No Intervention): Patients in this arm will not undergo one-hour application of abdominal Jackson-Pratt drain at the end of laparoscopic procedure.

INTERVENTIONS:
Device: abdominal Jackson-Pratt drain — One-hour application of abdominal Jackson-Pratt drain at the end of laparoscopic procedure.
  Arms: Abdominal Jackson-Pratt drain

SUMMARY:
Recent evidence has shown that the onset and intensity of post-operative pain are significantly related to the amount of residual pneumoperitoneum at the end of the surgical procedure. In addition, the use of low pressures of carbon dioxide (CO2) for induction of the pnemoperitoneum has been associated with a reduction in post-operative pain, probably due to a lower abdominal distension and a consequent reduced compression of the pelvic, abdominal and sub-diaphragmatic pain nerve fibers.

The reduction of the residual pnemoperitoneum at the end of the surgical procedure could therefore play a key role in the reduction of post-operative pain, with consequent greater comfort for the patient and reduction of the use of analgesics.

In view of the available evidence, the aim of the present study is to evaluate whether the application of Jackson-Pratt drain, for one hour from the end of the surgical procedure, can significantly reduce post-operative pain and the need of analgesics in patients undergoing laparoscopic gynecological surgery.

DETAILED DESCRIPTION:
Laparoscopy in gynecological surgery offers numerous advantages, such as the reduction of operative time, intra-operative blood loss, post-operative pain and the possibility of early hospital discharge and return to normal daily activities in a short time.

Despite these points arewidely validated in the literature, sometimes patients undergoing laparoscopy complain of abdominal pains (although slight in intensity and temporary) in the post-operative period. In some cases, the pain is characteristically irradiated at the shoulders, due to a probable irritation/compression of the phrenic nerve that runs on the lower surface of the diaphragm.

Recent evidence has shown that the onset and intensity of post-operative pain are significantly related to the amount of residual pneumoperitoneum at the end of the surgical procedure. In addition, the use of low pressures of carbon dioxide (CO2) for induction of the pnemoperitoneum has been associated with a reduction in post-operative pain, probably due to a lower abdominal distension and a consequent reduced compression of the pelvic, abdominal and sub-diaphragmatic pain nerve fibers.

The reduction of the residual pnemoperitoneum at the end of the surgical procedure could therefore play a key role in the reduction of post-operative pain, with consequent greater comfort for the patient and reduction of the use of analgesics.

In view of the available evidence, the aim of the present study is to evaluate whether the application of Jackson-Pratt drain, for one hour from the end of the surgical procedure, can significantly reduce post-operative pain and the need of analgesics in patients undergoing laparoscopic gynecological surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by uterine fibroids, undergoing laparoscopic surgery;
* American Society of Anesthesiologists physical status classification I-II.

Exclusion Criteria:

* inability to express pain;
* any concomitant diseases requiring upper abdominal surgery, such as cholecystectomy or adhesiolysis;
* laparoscopic procedures that were converted to open surgery;
* other causes of known pain;
* oncological cases;
* use of drugs for chronic pelvic pain or hormones in the previous 3 months (wash-out period);
* application of other drainages;
* intra- or post-operative complications.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Pain | 6 hours after surgery.
  Pain perception, expressed as Visual Analogue Score (0-10).

SECONDARY OUTCOMES:
Pain | 12 hours after surgery.
  Pain perception, expressed as Visual Analogue Score (0-10).
Pain | 24 hours after surgery.
  Pain perception, expressed as Visual Analogue Score (0-10).
Use of Analgesic | During the 48 hours after surgery.
  Number of requests for rescue analgesia (30 mg ketorolac tromethamine, administrated intravenously).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Insubria, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided